CLINICAL TRIAL: NCT06921837
Title: A Phase 1/2, First-in-Human, Dose Escalation and Expansion Study of BDC-4182 as a Single Agent in Patients With Advanced Gastric and Gastroesophageal Cancer
Brief Title: A First-in-Human Study Using BDC-4182 as a Single Agent in Advanced Gastric and Gastroesophageal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bolt Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BBI-4182-101
Record Dates: First submitted 2025-04-04; First posted 2025-04-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-11

CONDITIONS: Gastric Cancer Adenocarcinoma Metastatic; Gastroesophageal Adenocarcinoma
Keywords: Gastric Cancer; Gastroesophageal Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dose Escalation (Experimental): Escalating doses followed by backfill of selected doses
  Interventions: Drug: BDC-4182
- Dose Expansion (Experimental): Expansion at determined RP2D
  Interventions: Drug: BDC-4182

INTERVENTIONS:
Drug: BDC-4182 — Immune stimulating antibody conjugate (ISAC), consisting of an anti-claudin 18.2 monoclonal antibody conjugated to a TLR 7/8 dual agonist

SUMMARY:
A first-in-human study using BDC-4182 as a single agent in gastric and gastroesophageal cancers

DETAILED DESCRIPTION:
This is a dose escalation study designed to evaluate the safety and tolerability of BDC-4182 to establish the recommended Phase 2 dose (RP2D). Participants will be enrolled in each dose cohort until the maximum tolerated dose (MTD) is reached. Additional participants may be enrolled into backfill cohorts at dose levels that have been cleared to collect additional safety and tolerability data. Additional participants may be enrolled at the determined RP2D in an expansion portion of the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Has disease that is measurable by Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1.
* Subjects must have histologically/cytologically confirmed gastric or gastroesophageal cancer that is metastatic (Stage 4) or unresectable (Stage 3).
* Subjects must have received at least 1-2 prior lines of locally available standard therapies or must be intolerant of standard therapies.
* For subjects in escalation: If prior Claudin 18 IHC expression is known, the subject must have some degree of Claudin 18 expression as defined as Positive or have expression ≥ 1% of tumor cells IHC ≥ 2+. Consult with Medical Monitor as needed.
* Adequate organ function
* Agree to have a biopsy prior to enrollment, at acceptable risk in the judgement of the Investigator. If a biopsy is not safely accessible or clinically feasible, an adequate archival tumor sample must be submitted.

Key Exclusion Criteria:

* Known central nervous system (CNS) metastases except for disease that is asymptomatic, clinically stable, and has not required steroids for at least 14 days before starting study treatment.
* Cardiac disease, pulmonary disease, or hepatic disease
* Active infection
* History of inflammatory eye disease
* Residual toxicity from a previous treatment
* Any investigational agent or standard anti-cancer therapies within 28 days before starting study treatment or within 5 estimated elimination half-lives, whichever is shorter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) graded according to CTCAE v5.0 | approximately 2 years
  Escalation period
Incidence and nature of AEs considered by the Investigator or Sponsor to be clinically relevant, attributable to study treatment, and meeting dose-limiting toxicity (DLT) criteria | Up to 21 days
  Escalation period

SECONDARY OUTCOMES:
Objective response rate (ORR) according to RECIST v. 1.1 | approximately 4 years
  Escalation and expansion periods
Duration of Response (DOR) | approximately 4 years
  Escalation and expansion periods
Disease control rate (DCR) | approximately 4 years
  Escalation and expansion periods
Progression-free survival (PFS) | approximately 4 years
  Escalation and expansion periods
Best Overall Response (BOR) | approximately 4 years
  Escalation and expansion periods
Overall survival (OS) | approximately 4 years
  Escalation and expansion periods
PK (Cmax) of BDC-4182 | approximately 4 years
  Escalation and expansion periods
PK (Cmin) of BDC-4182 | approximately 4 years
  Escalation and expansion periods
PK (AUC0-tau) of BDC-4182 | approximately 4 years
  Escalation and expansion periods
PK (AUC0-inf) of BDC-4182 | approximately 4 years
  Escalation and expansion periods
PK (CL) of BDC-4182 | approximately 4 years
  Escalation and expansion periods
PK (Vc or Vss) of BDC-4182 | approximately 4 years
  Escalation and expansion periods
PK (Terminal half-life) of BDC-4182 | approximately 4 years
  Escalation and expansion periods

CONTACTS AND LOCATIONS:
Overall Officials: Bolt Clinical Development, Study Director — Bolt Biotherapeutics
Locations (16):
- Australia (5):
  - AUS Site 2, Darlinghurst, New South Wales
  - AUS Site 5, Westmead, New South Wales
  - AUS Site 1, Birtinya, Queensland
  - AUS Site 4, Clayton, Victoria
  - AUS Site 3, Heidelberg, Victoria
- South Korea (5):
  - SK Site 2003, Seongnam-si
  - SK Site 2001, Seoul
  - SK Site 2002, Seoul
  - SK Site 2004, Seoul
  - SK Site 2005, Seoul
- Taiwan (6):
  - TWN Site 9004, Kaohsiung City
  - TWN Site 9005, Kaohsiung City
  - TWN Site 9001, Taichung
  - TWN Site 9003, Taipei
  - TWN Site 9006, Taipei
  - TWN Site 9002, Taoyuan District

IPD SHARING:
Plan to Share IPD: No